CLINICAL TRIAL: NCT00392379
Title: Evaluating Nicotine Lozenges for Treatment of Smokeless Tobacco Addiction
Brief Title: Nicotine Lozenges for Treatment of Smokeless Tobacco Addiction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jon Ebbert, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-003091; R01CA121165 (NIH)
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2013-04

CONDITIONS: Smokeless Tobacco Use
Keywords: Tobacco use disorder; Tobacco cessation
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use Cessation | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): 4 mg nicotine lozenges for 3 months
  Interventions: Drug: Nicotine Lozenges
- B (Placebo Comparator): Placebo nicotine lozenges for 3 months
  Interventions: Drug: Placebo lozenge

INTERVENTIONS:
Drug: Nicotine Lozenges — Nicotine lozenges, 4 mg
  Other Names: Commit nicotine lozenge
  Arms: A
Drug: Placebo lozenge — Placebo lozenge
  Arms: B

SUMMARY:
This study will be a randomized, blinded, placebo-controlled two-group clinical trial. The independent variable is treatment assignment (active 4-mg nicotine lozenge vs. matching placebo lozenge), and the dependent variables are all tobacco and ST abstinence at 3 and 6 months. ST users will be randomly assigned to either the 4-mg active nicotine lozenge or matching placebo.

DETAILED DESCRIPTION:
Smokeless tobacco (ST) users will be randomly assigned to either the 4-mg active nicotine lozenge or matching placebo. Both groups will receive a behavioral intervention. The two sites for this clinical trial will be the Mayo Clinic in Rochester, Minnesota (central coordinating site) and the Oregon Research Institute (ORI) in Eugene, OR. A total of 270 ST users will be recruited into this clinical trail. All subjects will be randomized to 4 mg Nicotine Lozenges (taken ad lib) or matching placebo. They will be on study medication for 12 weeks and followed up for 6 months from study enrollment

ELIGIBILITY:
Inclusion Criteria:

* are at least 18 years of age;
* report smokeless tobacco (ST) as their primary tobacco of use;
* have used ST daily for the past 6 months;
* are in general good health (determined by medical history and screening physical examination);
* have been provided with, understand, and have signed the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon O. Ebbert, M.D., Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Oregon Research Institute, Eugene, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Mayo Clinic in Rochester, MN, and the Oregon Research Institute (ORI) in Eugene, OR. Enrollment took place between January, 2007 and April, 2008. Smokeless tobacco (ST) users were recruited through press releases and advertising from the surrounding communities.
Groups:
- Nicotine Lozenge; Placebo Nicotine Lozenge: Medication was given for 12 weeks. All subjects were instructed to quit all tobacco products and start using lozenges the following day. For weeks 1 through 6, subjects were instructed to use one lozenge orally every 1 to 2 hours with a maximum of 16 lozenges per day. After 6 weeks, lozenges were tapered. For weeks 7 through 9, subjects were instructed to use 8 lozenges per day or one every 2 to 4 hours. For weeks 10 through 12, subjects were instructed to use 4 lozenges per day or one every 4 to 8 hours.
Period: Overall Study
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge
Started | 136 (Medication period) | 134 (Medication period)
Completed | 114 (Medication period) | 96 (Medication period)
Not Completed | 22 | 38
Not completed — Withdrawal by Subject | 17 | 28
Not completed — Lost to Follow-up | 4 | 9
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge | Total
Number analyzed (Participants) | 136 | 134 | 270
Age Continuous [Mean (Standard Deviation); unit: years] | 36.6 (10.7) | 36.5 (11.0) | 36.6 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 136 | 128 | 264
Region of Enrollment [Number; unit: participants]
  United States | 136 | 134 | 270
ST Use [Mean (Standard Deviation); unit: Cans/week] — Can's week
  Cans/week | 4.3 (2.6) | 4.2 (2.6) | 4.2 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Smokeless Tobacco Abstinence at 3 Months
Description: Participants had to have self-reported not having used any tobacco from two weeks past the target quit date to the 3-months post baseline.
Time Frame: 3 months
Population: ITT
Measure: Number; unit: Participants
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge
Number analyzed (Participants) | 136 | 134
Participants | 65 | 41
Statistical Analysis 1: Comparison: Nicotine Lozenge vs Placebo Nicotine Lozenge; Based upon previous research, we hypothesized that the end-of-treatment abstinence rate for subjects receiving placebo would be 35% and the abstinence rate for subjects receiving the 4-mg nicotine lozenge would be 53%. A resulting power calculation indicated that 270 subjects (135 per group) were required in order to have 85% power to detect a significant difference (two-sided, α = 0.05 level test); Test type: Superiority or Other; p < 0.05, Regression, Logistic — No adjustment for multiple comparisons; Odds Ratio (OR) = 3, Standard Deviation 43

2. Secondary Outcome: Self-reported Point Prevalence All Tobacco Abstinence at 3 Months
Description: Participants had to have self-reported not having used any tobacco for the 7 days prior to the 3 month visit.
Time Frame: 3 months
Measure: Number; unit: Participants
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge
Number analyzed (Participants) | 136 | 134
Participants | 60 | 39

3. Secondary Outcome: Prolonged Smokeless Tobacco Abstinence at 6 Months
Description: Participants had to have self-reported not having used any tobacco from 2 weeks after the target quit date to 6 months after baseline (22 weeks).
Time Frame: 6 months
Measure: Number; unit: Participants
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge
Number analyzed (Participants) | 136 | 134
Participants | 41 | 31

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Nicotine Lozenge | Placebo Nicotine Lozenge
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/134
Other Adverse Events (participants affected / at risk) | 33/136 | 17/134
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine Lozenge (N=136) | Placebo Nicotine Lozenge (N=134)
Reflux (Gastrointestinal disorders) | 15 | 1
Sleep disturbance (Nervous system disorders) | 8 | 9
Headache (Nervous system disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No